CLINICAL TRIAL: NCT03326700
Title: Effects of Laparoscopic Totally Extraperitoneal and Lichtenstein Hernia Repair on Men's Sexual Functions and Quality of Life.
Brief Title: Effects of Hernia Repair on Men's Sexual Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Riza Gurhan ISIL, MD, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEEAH 2015 / 568
Record Dates: First submitted 2017-10-22; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Hernia, Inguinal; Men; Sexual Dysfunction
MeSH Terms: conditions — Hernia, Inguinal; Multiple Endocrine Neoplasia Type 1; Sexual Dysfunction, Physiological

STUDY DESIGN:
Intervention Model Description: 176 men with unilateral inguinal hernia were randomized in two groups. Group T(n=88) were operated TEP and Group L(n:88) were operated by LH repair. Patients demografigs, perioperative findings were recorded. For all patients preoperative, postoperative 7th,30th and 90th day SF 36 and IIEF were filled up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic hernia repair. (Active Comparator): Intervention: inguinal hernia repair.
  Interventions: Procedure: Inguinal Hernia Repair
- Open hernia repair. (Active Comparator): Intervention: inguinal hernia repair.
  Interventions: Procedure: Inguinal Hernia Repair

INTERVENTIONS:
Procedure: Inguinal Hernia Repair — Inguinal hernia repair is surgery to repair a hernia in the groin. A hernia is tissue that bulges out of a weak spot in the abdominal wall. The intestine may bulge out through this weakened area. During surgery to repair the hernia, the bulging tissue is pushed back in. The abdominal wall is strengthened and supported with sutures (stitches), and sometimes mesh. This repair can be done with open or laparoscopic surgery.

SUMMARY:
In the literature, there are several studies that compare Laparoscopic totally extraperitoneal hernia repair (TEP) with Lichtenstein hernia (LH) repair. There are no studies that compare sexual functions on men's health and quality of life. Our aim was to study the sexual functions of men, who underwent TEP or LH repair according to Health Survey Scoring Demonstration (SF36) and The International Index of Erectile Function (IIEF).

DETAILED DESCRIPTION:
176 men with unilateral inguinal hernia were randomized into two groups. Group T (n=88) underwent TEP and Group L(n:88) underwent LH repair. Patients demografigs, perioperative findings were recorded. For all patients preoperative, postoperative 7th,30th and 90th day SF 36 and IIEF were filled up.

ELIGIBILITY:
Inclusion Criteria:

* having male gender
* patients diagnosed on unilateral inguinal hernia
* patients aged between 18 and 65 years
* ASA I and II patients

Exclusion Criteria:

* having female gender
* patients diagnosed on bilateral or recurrence inguinal hernia,
* patients suffering erectile dysfunction

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
IIEF Scale | 7 to 90 days
  international index of erectile functions

SECONDARY OUTCOMES:
SF36 | 7 to 90 days
  health survey scoring demonstration

IPD SHARING:
Plan to Share IPD: No
We can share study data only without patients names.

REFERENCES:
- [Background] Kushwaha JK, Enny LE, Anand A, Sonkar AA, Kumar A, Pahwa HS. A Prospective Randomized Controlled Trial Comparing Quality of Life Following Endoscopic Totally Extraperitoneal (TEP) Versus Open Stoppa Inguinal Hernioplasty. Surg Laparosc Endosc Percutan Tech. 2017 Aug;27(4):257-261. doi: 10.1097/SLE.0000000000000450. PMID 28727632